CLINICAL TRIAL: NCT04168892
Title: Prospective, Observational, Multivariate Study to Evaluate the Best Predictor of Ovarian Response, Between AMH Measured With Fully Automated Assay and AFC
Brief Title: Anti-Müllerian Hormone (AMH) Measured With Fully Automated Assay Versus AFC in the Prediction of Ovarian Response
Status: Completed | Type: Observational
Sponsor: Andros Day Surgery Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 01/MR/19
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Ovarian Response
MeSH Terms: interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female age ≤ 35 years: 150 IU of HMG: For controlling the effect of the starting dose on the number of retrieved oocytes, the patients will be divided in two groups based on their age. For the patients with an age ≤ 35 years, COS will be carried out by daily injections of 150 IU of Human Menopausal Gonadotropins (HMG) and will be started on the 3rd day of the cycle. The starting dose will be maintained for the first 5 days and followed by individual dose-adjustments according to the patient's follicular response. The pituitary suppression will be obtained by the administration of the Gonadotropin-releasing Hormone (GnRH) antagonist ganirelix (0.25 mg per day), starting from the 6th day of the ovarian stimulation until the day of the induction of the final oocyte maturation. Highly purified urinary human Chorionic Gonadotropin (hCG) 10.000 IU will be used to induce final oocyte maturation. In case of OHSS risk, the final oocyte maturation will be obtained by using a GnRH agonist (buserelin acetate), 0.5 mg subcutaneously.
  Interventions: Drug: 150 IU of HMG in patients with age ≤ 35 years
- Female age >35 years: 225 IU of HMG: In order to control the effect of the starting dose on the number of retrieved oocytes, the patients will be divided in two groups based on their age. For the patients with an age >35 years, the controlled ovarian stimulation will be carried out by daily injections of 225 IU of HMG and will be started on the 3rd day of the cycle. The starting dose will be maintained for the first 5 days and followed by individual dose-adjustments according to the patient's follicular response. The pituitary suppression will be obtained by the administration of the GnRH antagonist ganirelix (0.25 mg per day), starting from the 6th day of the ovarian stimulation until the day of the induction of the final oocyte maturation. Highly purified urinary hCG 10.000 IU will be used to induce final oocyte maturation. In case of OHSS risk, the final oocyte maturation will be obtained by using a GnRH agonist (buserelin acetate), 0.5 mg subcutaneously.
  Interventions: Drug: 225 IU of HMG in patients with age > 35 years

INTERVENTIONS:
Drug: 150 IU of HMG in patients with age ≤ 35 years — The use of a different starting dose, based on the female age, derives from the necessity to control the effect of a variable starting dose on the primary outcome.
  Groups: Female age ≤ 35 years: 150 IU of HMG
Drug: 225 IU of HMG in patients with age > 35 years — The use of a different starting dose, based on the female age, derives from the necessity to control the effect of a variable starting dose on the primary outcome.
  Groups: Female age >35 years: 225 IU of HMG

SUMMARY:
The primary objective of this prospective, observational, multivariate study will be to compare the reliability of automated AMH (measured with Access AMH assay, Beckman-Coulter Diagnostics, USA) with that of antral follicle count (AFC) evaluated ultrasonographically always by the same operator and with the same ultrasound scanner, in terms of the number of oocytes recovered from oocyte sampling in couples subjected to in vitro fertilization.

DETAILED DESCRIPTION:
Individual variability in ovarian response to a starting dose of gonadotropins is a well-known aspect during controlled ovarian stimulation (COS) and many efforts have been made for obtaining the personalization of the treatment, identifying different biomarkers that may predict the ovarian response such as age, basal Follicle Stimulating Hormone (FSH), AMH and antral follicle count (AFC). The number of oocytes retrieved is the main expression of ovarian response and it remains a relevant prognostic marker in women undergoing In Vitro Fertilization (IVF)/Intracytoplasmic Sperm Injection (ICSI) cycles. Consistent evidence shows that an optimal - rather than a maximal - oocyte yield is the preferred achievement after COS when fresh embryo transfer is scheduled. In fact, live birth rates steadily increase when an optimal number of oocytes is collected, whereas low response and hyper-response are associated with lower implantation rates, increased obstetrical risks and, at least when considering hyper response, increased risk of ovarian hyperstimulation syndrome (OHSS) in the fresh cycle. Among the different biomarkers, AMH and AFC seem to have the best performance in predicting ovarian response to exogenous FSH.

Nevertheless, until now, there is often discordance between the AMH level and AFC in clinical practice. In cases of discordance, which indicator should be chosen to individualize the starting dose of gonadotropins? Until now, no direct comparison of the new automated immunoassay of AMH with AFC has been carried out considering the number of retrieved oocytes as primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

BMI between 18 and 30 kg/m2, basal serum day 3 FSH ≤ 15 IU/l, normal regular menstrual cycles, ranging from 25 to 33 days in length, normal thyroid-stimulating hormone (TSH) and prolactin levels, normal uterine cavity as assessed by hysteroscopy or sonohysterography or three-dimensional ultrasound and presence of both ovaries.

Exclusion Criteria:

irregular menstrual cycles, severe endometriosis, defined as stage III-IV of the American Society for Reproductive Medicine (ASRM) revised classification, previous ovarian surgery, presence of ovarian cysts, polycystic ovary syndrome, use of hormonal contraception in the previous 3 months and use of gonadotrophins in the previous 3 months, any known metabolic or endocrinological disease

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: This trial will involve couples attending their first IVF/ICSI cycle.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 13-15 days starting from the first day of the cycle
  The number of oocytes collected after oocyte retrieval

SECONDARY OUTCOMES:
Cumulative clinical pregnancy rate per patient | 28-32 days after the oocyte retrieval
  The number of clinical pregnancies (gestational sacs with a fetal heartbeat detected at ultrasound 28-32 days after oocyte retrieval) obtained by fresh and frozen embryo transfers per each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- ANDROS Day Surgery Clinic, Reproductive Medicine Unit, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Xu Y, Xue Q, Shang J, Yang X, Shan X, Kuai Y, Wang S, Zeng C. Discordance between antral follicle counts and anti-Mullerian hormone levels in women undergoing in vitro fertilization. Reprod Biol Endocrinol. 2019 Jul 4;17(1):51. doi: 10.1186/s12958-019-0497-4. PMID 31272468
- [Background] Pearson K, Long M, Prasad J, Wu YY, Bonifacio M. Assessment of the Access AMH assay as an automated, high-performance replacement for the AMH Generation II manual ELISA. Reprod Biol Endocrinol. 2016 Feb 16;14:8. doi: 10.1186/s12958-016-0143-3. PMID 26879773
- [Background] Allegra A, Marino A, Volpes A, Coffaro F, Scaglione P, Gullo S, La Marca A. A randomized controlled trial investigating the use of a predictive nomogram for the selection of the FSH starting dose in IVF/ICSI cycles. Reprod Biomed Online. 2017 Apr;34(4):429-438. doi: 10.1016/j.rbmo.2017.01.012. Epub 2017 Jan 23. PMID 28189417
- [Background] van Tilborg TC, Oudshoorn SC, Eijkemans MJC, Mochtar MH, van Golde RJT, Hoek A, Kuchenbecker WKH, Fleischer K, de Bruin JP, Groen H, van Wely M, Lambalk CB, Laven JSE, Mol BWJ, Broekmans FJM, Torrance HL; OPTIMIST study group. Individualized FSH dosing based on ovarian reserve testing in women starting IVF/ICSI: a multicentre trial and cost-effectiveness analysis. Hum Reprod. 2017 Dec 1;32(12):2485-2495. doi: 10.1093/humrep/dex321. PMID 29121350
- [Background] Andersen AN, Witjes H, Gordon K, Mannaerts B; Xpect investigators. Predictive factors of ovarian response and clinical outcome after IVF/ICSI following a rFSH/GnRH antagonist protocol with or without oral contraceptive pre-treatment. Hum Reprod. 2011 Dec;26(12):3413-23. doi: 10.1093/humrep/der318. Epub 2011 Sep 27. PMID 21954280